CLINICAL TRIAL: NCT06870331
Title: The Effect of Probiotic and Prebiotic Supplementation on Gastrointestinal Health in Individuals With Chronic Spinal Cord Injury: A Randomized Controlled Crossover Trial
Brief Title: The Effect of Probiotic and Prebiotic Supplementation on Gastrointestinal Health in Individuals With Chronic Spinal Cord Injury
Acronym: PRO-GIDSCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024-25
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injury
Keywords: probiotic; prebiotic; gastrointestinal health; microbiome; dietary supplement
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Probiotics; Prebiotics

STUDY DESIGN:
Intervention Model Description: Open-label two-arm randomized controlled crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic intervention (Experimental): Probiotics add beneficial bacterial strains to the gut, which can restore microbial balance.
  Interventions: Dietary Supplement: Probiotic
- Prebiotic intervention (Active Comparator): Prebiotics, such as oat bran, selectively promote the growth of beneficial gut bacteria, particularly butyrate-producing species.
  Interventions: Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants will take one sachet BIOTICS-G (Burgerstein, Switzerland, 2.5 g) daily for eight weeks. The supplement contains 14 bacterial strains with a total viable cell count of 2.5 billion colony-forming units per sachet.
  Arms: Probiotic intervention
Dietary Supplement: Prebiotic — Participants will take 5 g of oat bran (Naturaplan Bio Haferkleie, Coop, Switzerland) daily for eight weeks.
  Arms: Prebiotic intervention

SUMMARY:
The goal of this clinical trial is to evaluate the effect of probiotic and prebiotic supplementation in individuals with chronic spinal cord injury experiencing gastrointestinal complaints.

The main questions this trail aims to answer are:

* what are the effects of the supplementation on gastrointestinal symptoms?
* what are the effects of the supplementation on gut microbiome composition?
* what are the effects of the supplementation on inflammatory serum markers?
* what are the effects of the supplementation on gastrointestinal transit time?

Participants will:

* take either the probiotic or prebiotic supplement daily for eight weeks, followed by a four-week "wash-out period" (= no intake of either supplement) and a subsequent eight-week intake of the other supplement.
* visit the study center for four appointments, during which various measurements will be performed.

ELIGIBILITY:
Inclusion Criteria (at screening):

* Age: ≥ 18 years
* Sex: male and female.
* Chronic SCI (>1 year post-injury)
* Individuals with para- and tetraplegia (American Spinal Cord Injury (ASIA) Impairment Scale (AIS) score A-D)
* Having significant gastrointestinal complaints, indicated with "yes" at screening and by a GIQLI questionnaire score below 110 at baseline
* Signed written informed consent

Exclusion Criteria (at screening):

* Antibiotic use within the last four weeks before starting the study
* Major dietary changes within the last four weeks before starting the study, such as initiating a vegan or ketogenic diet
* Presence of clinically relevant medical conditions, including Crohn's disease, diagnosed eating or gastrointestinal disorders, assessed on an individual basis
* Intake of significant concomitant medication, including immunomodulating therapy, mesalazines, or steroids, assessed on an individual basis
* Concurrent participation in other clinical trials investigating or potentially affecting GI health
* Insufficient German language skills to follow the study procedures
* Pregnancy (anamnestic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | Before and after eight weeks of intake of the dietary supplement.
  Change in gastrointestinal symptoms using the Gastrointestinal Quality of Life (GIQLI) questionnaire.

SECONDARY OUTCOMES:
Gut microbiome composition | Before and after eight weeks of intake of the dietary supplement.
  Change in gut microbiome composition, assessed using a stool sample.
Inflammatory markers | Before and after eight weeks of intake of the dietary supplement.
  Change in serum inflammatory markers, assessed by a blood sample.
Gastrointestinal transit time | Before and after eight weeks of intake of the dietary supplement.
  Change in gastrointestinal transit time, assessed by the blue dye test (time from ingestion to first appearance of blue food dye in the stool).

OTHER OUTCOMES:
Side effects | After the eight weeks of intake of the dietary supplement.
  Occurrence of side effects of the supplementation, assessed by questioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jivko Stoyanov, Prof. Dr., Study Director — Swiss Paraplegic Research, Nottwil
Locations (1):
- Swiss Paraplegic Research, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trunz J, Schmandt C, Hertig-Godeschalk A, Glisic M, Stoyanov J, Perret C. Probiotic and Prebiotic Supplementation for Gastrointestinal Discomfort in Chronic Spinal Cord Injury (PRO-GIDSCI): A Randomized Controlled Crossover Trial Protocol. Methods Protoc. 2026 Jan 17;9(1):14. doi: 10.3390/mps9010014. PMID 41562992